CLINICAL TRIAL: NCT00720369
Title: Oral Administration of CoQ10 and Phosphorus-31 Magnetization Transfer Magnetic Resonance Spectroscopy in Geriatric Bipolar Disorder and Healthy Older Adults
Brief Title: CoQ10 in Geriatric Bipolar Depression
Acronym: CoQ10
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, Brent Forester, Director, Mood Disorders Division, Geriatric Psychiatry Research Program, Mclean Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2008-P-000738/1
Record Dates: First submitted 2008-07-18; First posted 2008-07-22 (Estimated); Results first posted 2014-01-13 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2013-11

CONDITIONS: Bipolar Depression
Keywords: Bipolar depression; elderly; Coenzyme Q10; Magnetic resonance spectroscopy
MeSH Terms: conditions — Bipolar Disorder | interventions — coenzyme Q10

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CoEnzyme Q10 (Experimental): Open Label Study
  Interventions: Drug: CoEnzyme Q10
- Healthy Controls (No Intervention): Healthy controls completed all study procedures completed by the CoQ10 group but did not receive any study medication.

INTERVENTIONS:
Drug: CoEnzyme Q10 — CoEnzyme Q10 with dosage range from 400 mg to 1200 mg per day
  Arms: CoEnzyme Q10

SUMMARY:
We propose to study and compare measures of brain energy metabolism in geriatric bipolar individuals and healthy older adults. We would also like to investigate changes in brain energy metabolites and in vivo creatine kinase (CK) enzymatic activity associated with CoQ10 administration in older bipolar individuals.

DETAILED DESCRIPTION:
Hypotheses

1. At baseline, the forward rate constant (kfor) of CK enzymatic activity in the frontal lobe of older subjects with bipolar depression will be significantly decreased relative to that of age-matched healthy controls.
2. After 8 weeks of treatment, bipolar depression subjects will demonstrate an increase in the kfor of CK after 8 weeks of CoQ 10 treatment.
3. Increases in the CK forward rate constant (kfor) will correlate with improvement in subjects' mood state as assessed by the Montgomery Asberg Depression Rating Scale (MADRS).
4. Baseline measures of executive functioning and information processing speed (measured by performance on the Wisconsin Card Sorting Test (WCST), Trails A and B and Stroop tests) will be impaired in subjects with geriatric bipolar depression compared with healthy controls. These measures will improve with successful treatment with CoQ10 and correlate with increases in the CK forward rate constant (kfor).

Summary:

A review of literature suggests a distinct pattern of bioenergetic changes, possibly related to mitochondrial dysfunction and abnormal CK function, in older adults and in individuals with bipolar disorder. As opposed to rudimentary measurements of static metabolite concentrations, the novel use of MT-MRS in such individuals will offer insight into the enzyme kinetics of CK, specifically examining the rate at which ATP is formed from PCr. From previous investigations it would seem that the dietary-supplement, CoQ10, is able to improve the efficiency of mitochondrial function in subjects with altered bioenergetics. We propose to measure CK activity and PCr turnover rate before and after CoQ10 treatment, with the overall aim of understanding metabolic relationships between brain bioenergetic alterations and treatment with CoQ10 in geriatric bipolar depression.

ELIGIBILITY:
Inclusion Criteria:

* 55 years or older
* Meet DSM-IV diagnostic criteria for Bipolar Disorder, Current Episode Depressed
* Montgomery Asberg Depression Rating Scale (MADRS) Score of >20
* If the MADRS score is <20 but >16, a diagnosis of bipolar disorder, current episode depressed, based on the Structured Clinical Interview of DSM IV TR (SCID) and Dr. Forester's initial interview would allow the subject to be included in the study.
* Young Mania Rating Scale (YMRS) Score of < 6
* If the YMRS score is >6 subjects can still be admitted if subjects do not meet clinical criteria for mania or hypomania at the time of screening
* Able to provide informed consent
* Must speak English
* Must be able to visit McLean Hospital for the screening visit and six study visits during the 8-week duration of the study
* Subjects may be taking other medications for bipolar depression including antidepressants, mood stabilizers and antipsychotic mediations prior to Co-Q10 therapy, but may not have any dosage adjustments of these medications in the week before Co-Q10 is added.

Exclusion Criteria:

* Serious or unstable medical illness, including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic or hematologic disease
* History of seizure disorder,
* History or current diagnosis of the following psychiatric illnesses: any organic mental disorder (including dementia), schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorder not otherwise specified, unipolar major depressive disorder, patients with substance dependence disorders, including alcohol, active within the last 12 months.
* History of drug hypersensitivity or intolerance to Coenzyme Q10.
* Use of medications that are excluded in this study (barbiturates; however, the use of non-benzodiazepine sedative hypnotics (such as zolpidem (Ambien)) may be used as needed except within 12 hours of the MRI scan)
* Benzodiazepines may be used by subjects throughout the study as long as they are not taken within 12 hours of any MRI scan.
* Subjects diagnosed with a mitochondrial disorder.
* Subjects taking other putative mitochondrial enhancers (e.g., vitamin E, carnitine, creatine, Vitamin complex B, pramipexole) at the time of study entry.
* Any of the exclusion criteria mentioned in the MRI risks section below

Ages: 55 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brent P Forester, MD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Please note that subjects who sign the informed consent form are considered "enrolled." Only subjects who met eligibility following screening are included in analyses and thus included in the "participant flow." Of the 42 enrolled, 19 started the study and 18 completed.
Groups:
- CoQ10: Subjects were given open-label, adjunct treatment with CoQ10 with oral dosing between 400-1200mg per day. Dosing was started at 400mg and titrated up to 1200mg as tolerated. This value does not match the value of subjects enrolled because only subjects who were not screen failures are included in this group.
- Healthy Controls: Healthy age matched control subjects do not receive treatment. Controls undergo testing and MRIs to serve as comparison group. This value does not match the value of subjects enrolled because only subjects who were not screen failures are included in this group.
Period: Overall Study
Arm/Group | CoQ10 | Healthy Controls
Started | 11 | 8
Completed | 10 (one subject discontinued due to an adverse event.) | 8
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CoQ10 | Healthy Controls | Total
Number analyzed (Participants) | 11 | 8 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 5 | 13
  >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (7.5) | 66.4 (9.5) | 64.6 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 11 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: We Measured the Change in Rate Constant of Creatine Kinase in Individuals With Bipolar Depression Treated With CoQ 10 as Compared With Age and Gender Matched Controls. These Rate Constants Were Calculated Using Magnetic Resonance Imaging (MRI).
Description: The rate constant for creatine kinase is a measurement of the reaction rate ADP+PCr <---> ATP + Cr, which is catalyzed by the enzyme creatine kinase. The rate constant shows the direction and magnitude of the reaction at equilibrium. A higher rate constant indicates a higher rate constant of the CK enzyme, meaning, more efficient/rapid conversion of PCr to ATP through the creatine kinase enzymatic reaction in tissues with high and fluctuating energy demands such as brain and muscle tissue. As the value is a reaction rate, there are no associated units.
Time Frame: 8 week trial
Measure: Mean (Standard Deviation); unit: per second
Groups:
- CoQ10: Subjects were given open-label, adjunct treatment with CoQ10 with oral dosing between 400-1200mg per day. Dosing was started at 400mg and titrated up to 1200mg as tolerated.
- Healthy Controls: Healthy age matched control subjects do not receive treatment. Controls undergo testing and MRIs to serve as comparison group.
Arm/Group | CoQ10 | Healthy Controls
Number analyzed (Participants) | 10 | 8
per second | 0.02 (0.002) | 0.03 (0.05)

2. Secondary Outcome: We Measured Response to Treatment of Depression (Using the Montgomery Asberg Depression Rating Scale)in Older Adults With Bipolar Disorder After an 8 Week Trial of CoQ10.
Description: The Montgomery Asberg Depression Rating Scale (MADRS) is a 10 question questionnaire which assesses symptom severity of depression. The score is on a 0-60 scale with higher numbers indicating more severe depressive symptoms. The score is represented as a number of points.
  Clinical improvement following treatment with CoQ10 supplement was only tested in the Bipolar subject cohort, not in healthy controls, therefore outcome data only apply to the bipolar group.
Time Frame: 8 week trial
Population: Clinical improvement following treatment with CoQ10 supplement was only tested in the Bipolar subject cohort, not in healthy controls, therefore outcome data only apply to the bipolar group.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- CoQ10: Open Label Study
- Healthy Controls: Clinical improvement following treatment with CoQ10 supplement was only tested in the Bipolar subject cohort, not in healthy controls, therefore outcome data only apply to the bipolar group.
Arm/Group | CoQ10 | Healthy Controls
Number analyzed (Participants) | 10 | 0
units on a scale
  Pre-Treatment (baseline) | 21.4 (5.5) |
  Post-Treatment (week 8) | 18.4 (7.3) |

ADVERSE EVENTS:
Arm/Group | CoQ10 | Healthy Controls
Serious Adverse Events (participants affected / at risk) | 0/11 | 1/8
Other Adverse Events (participants affected / at risk) | 9/11 | 2/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CoQ10 (N=11) | Healthy Controls (N=8)
chest pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Subject admitted to ER with chest pain, diagnosed with pneumonia, deemed to be unrelated to study participation by PI.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CoQ10 (N=11) | Healthy Controls (N=8)
discomfort in MRI (General disorders) | 0 (0) | 1 (1)
flu like symptoms (Infections and infestations) | 0 (0) | 1 (1)
fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
persistence of pre-existing atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
hair loss (General disorders) | 1 (1) | 0 (0)
eye pain (Eye disorders) | 1 (2) | 0 (0)
headache (Nervous system disorders) | 2 (2) | 0 (0)
dizziness (Nervous system disorders) | 1 (1) | 0 (0)
food poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No